CLINICAL TRIAL: NCT06205693
Title: Intraoperative Biodegradable Stent Placement to Reduce Complications After Pancreatoduodenectomy - Protocol and Statistical Analysis Plan for Randomized, Clinical Trial
Brief Title: Intraoperative Biodegradable Stent Placement to Reduce Complications After Pancreatoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Waqas Farooqui, Generel Surgeon, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Stent-trial
Record Dates: First submitted 2023-12-14; First posted 2024-01-16 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Fistula Pancreatic
Keywords: Fistula; postoperative pancreatic fistula; pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula; Fistula

STUDY DESIGN:
Intervention Model Description: prospective, randomized, blinded clinical superiority trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigators will mask the allocation for the outcome assessors and trial statistician who will conduct the analyses, and the author group while writing the abstract for the trial report with the two intervention groups coded as 0 and 1. Due to the nature of the intervention and control, the trial will not be blinded for the surgeons performing the interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stent (Active Comparator): Placement of biodegradable stent intraoperatively.
  Interventions: Procedure: Fast Degradable, Biodegradable ARCHEMEDES stent
- No stent (No Intervention): Control group. No placement of stent.

INTERVENTIONS:
Procedure: Fast Degradable, Biodegradable ARCHEMEDES stent — Fast Degradable, Biodegradable ARCHEMEDES stent. Placed in the pancreaticojejunostomy.
  Arms: Stent

SUMMARY:
The aim of this prospective, randomized, blinded clinical superiority trial is to establish intraoperative placement of biodegradable stents in the pancreatojejunostomy as a safe, effective, and feasible preventive measure against pancreatic fistula following pancreatoduodenectomy.

The investigators hypothesize that intraoperative placement of biodegradable stents in the pancreatojejunostomy is safe and can reduce the risk of pancreatic leakage following pancreatoduodenectomy in patients who have not undergone PBD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing a pancreatoduodenectomy
2. Patients aged 18 or above
3. Patients who have given an informed consent

Exclusion Criteria:

1. Patients who do not or cannot give an informed consent.
2. Patients with at a high risk or with previous history of multiple thrombo-embolic diseases or bleeding disorders.
3. Patients undergoing active immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
POPF | 30 days
  Number of participants with a Postoperative pancreatic fistula
Number of participants with a Biliary fistula | 30 days
  Postoperative biliary fistula

SECONDARY OUTCOMES:
Complications to stent placement | 30 days
  Incidence of complications to placement of the biodegradable stent, including displacement.
Postoperative complications | 30 days postoperative
  Overall incidence of complications following PD classified according to Clavien-Dindo
Mortality | 30 days and 90 days
  Participant Mortality at 30 and 90 days
LOS | Length in days, from surgery until discharge ( up to 200 days from surgery)
  Participant Length of hospital stay (LOS).
Quality of Life according to VR12 Quality of Life Score | 30 days post surgery
  Patient reported quality of life according to VR12 Quality of Life Score (activity level, pain episodes, pain levels, patient mood)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Capitol, Denmark

IPD SHARING:
Plan to Share IPD: Undecided